CLINICAL TRIAL: NCT03485105
Title: Prediction of Benefit From Adjuvant Chemotherapy for pT1N1 Gastric Cancer: A Pilot Retrospective Multicenter Cohort Study
Brief Title: Prediction of Benefit From Adjuvant Chemotherapy for pT1N1 Gastric Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2017-0914
Record Dates: First submitted 2018-03-26; First posted 2018-04-02 (Actual); Last update posted 2018-04-09 (Actual); Status verified 2018-03

CONDITIONS: Gastric Cancer
Keywords: Gastric cancer; biomarker; chemotherapy; precise medicine
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — specimen including mRNA from formalin fixed paraffin embeded tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- CTX-benefit group: CTX-benefit group: based on the result of nProfiler Stomach cancer assay kit which was decided by expression level of mRNA, this group will be beneficial from adjuvant chemotherapy
- no-benefit group: no-benefit group: based on the result of nProfiler Stomach cancer assay kit which was decided by expression level of mRNA, this group will not be beneficial from adjuvant chemotherapy
- high-risk group: high-risk group: based on the result of nProfiler Stomach cancer assay kit which was decided by expression level of mRNA, the prognosis of this group will be worse compared to others regardless of the response to adjuvant chemotherapy

SUMMARY:
To conduct a retrospective study to prove a hypothesis of "adjuvant chemotherapy provides survival benefit for patients of CTX-benefit group in gastric cancer of pT1N1, especially in high-risk group". This study is a pilot study and the result will be used as a reference for the upcoming prospective randomized controlled trial for same issue including estimating sample size. Two high-volume hospitals (Yonsei University Severance Hospital and Samsung Hospital) will participant this pilot study.

FFPE sample blocks and clinical information pertaining to the patients who satisfied with selection criteria will be collected from two institutions. The primary end point of this study is disease-free survival (DFS) that is defined as the time from surgery to death or gastric cancer recurrence whichever occurred first; and overall survival (OS) that is defined as time from surgery to death by any causes. Clinical information such as age, sex, histology, Lauren classification, depth of invasion, number of retrieved and metastatic lymph nodes, sizes of tumor, location of tumor, gross type, lympho-vascular invasion, received chemotherapy or not will be centralized.

One or 2 of 3mm core of tumor will be punched from FFPE and it will be delivered through Eppendorf tube to laboratory (Novomics Co. Ltd., Seoul, Korea). RNA will be extracted from the tissue and the pattern of RNA expression will be evaluated and each sample will be categorized into three risk group (high, intermediate, low risk group) and two predictive group (CTX-benefit and no-benefit group) by GMP-grade nProfiler 1TM Stomach Cancer Assay Kit (Novomics Co. Ltd., Seoul, Korea). Both clinical information and classification will be delivered to independent statisticians who are responsible to conduct statistical analyses.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed gastric adenocarcinoma
2. Patients who received R0 resection with curative intent surgery
3. pT1 (mucosa/submucosa) N1(one or two metastatic lymph nodes) M0
4. patients received surgery with lymph node dissection of D1 + or more
5. number of retrieved lymph nodes >15
6. Formalin-Fixed Paraffin-Embedded cancer tissues are available
7. Adults over 19 years

Exclusion Criteria:

1. Patients received pre-operative chemotherapy or radiotherapy
2. Cancer in remnant stomach (history of gastrectomy)
3. in hospital mortality or died within 30 days after surgery
4. FFPE is not available

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: approximately 1,000 patients Formalin-fixed, paraffin-embedded (FFPE) sample blocks from patients who treated at Severance Hospital and Samsung Hospital for gastric cancer (satisfied with below criteria) with pT1N1 stage and their corresponding clinical information will be evaluated from 1990-2012, approximately 500 participants in each hospital).
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-10-01 (Estimated); Study Completion 2019-11-01 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | average 5 years to detect recurrence of tumor
  Disease free survival which is defined as the time from surgery to death or gastric cancer recurrence whichever occurred first, and overall survival that is defined as time from surgery to death by any causes
overall survival | average of follow up duration will be 60 months
  overall survival that is defined as time from surgery to death by any causes. Survival difference between surgery only vs. surgery plus adjuvant treatment (chemotherapy or chemo-radiotherapy) will be analyzed according to subgroup (CTX-benefit and no-benefit group in overall and high-risk group)

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Upper Gastrointestinal Surgery, Department of Surgery, Yonsei University College of Medicine, Seoul, South Korea

REFERENCES:
- [Background] Cheong JH, Yang HK, Kim H, Kim WH, Kim YW, Kook MC, Park YK, Kim HH, Lee HS, Lee KH, Gu MJ, Kim HY, Lee J, Choi SH, Hong S, Kim JW, Choi YY, Hyung WJ, Jang E, Kim H, Huh YM, Noh SH. Predictive test for chemotherapy response in resectable gastric cancer: a multi-cohort, retrospective analysis. Lancet Oncol. 2018 May;19(5):629-638. doi: 10.1016/S1470-2045(18)30108-6. Epub 2018 Mar 19. PMID 29567071
- [Background] Nakajima T, Nashimoto A, Kitamura M, Kito T, Iwanaga T, Okabayashi K, Goto M. Adjuvant mitomycin and fluorouracil followed by oral uracil plus tegafur in serosa-negative gastric cancer: a randomised trial. Gastric Cancer Surgical Study Group. Lancet. 1999 Jul 24;354(9175):273-7. doi: 10.1016/s0140-6736(99)01048-x. PMID 10440302
- [Background] Shin HB, An JY, Lee SH, Choi YY, Kim JW, Sohn SS, Noh SH. Is adjuvant chemotherapy necessary in pT1N1 gastric cancer? BMC Cancer. 2017 Apr 22;17(1):287. doi: 10.1186/s12885-017-3265-x. PMID 28431518
- [Background] Noh SH, Park SR, Yang HK, Chung HC, Chung IJ, Kim SW, Kim HH, Choi JH, Kim HK, Yu W, Lee JI, Shin DB, Ji J, Chen JS, Lim Y, Ha S, Bang YJ; CLASSIC trial investigators. Adjuvant capecitabine plus oxaliplatin for gastric cancer after D2 gastrectomy (CLASSIC): 5-year follow-up of an open-label, randomised phase 3 trial. Lancet Oncol. 2014 Nov;15(12):1389-96. doi: 10.1016/S1470-2045(14)70473-5. Epub 2014 Oct 15. PMID 25439693
- [Background] Sasako M, Sakuramoto S, Katai H, Kinoshita T, Furukawa H, Yamaguchi T, Nashimoto A, Fujii M, Nakajima T, Ohashi Y. Five-year outcomes of a randomized phase III trial comparing adjuvant chemotherapy with S-1 versus surgery alone in stage II or III gastric cancer. J Clin Oncol. 2011 Nov 20;29(33):4387-93. doi: 10.1200/JCO.2011.36.5908. Epub 2011 Oct 17. PMID 22010012
- [Background] Japanese Gastric Cancer Association. Japanese classification of gastric carcinoma: 3rd English edition. Gastric Cancer. 2011 Jun;14(2):101-12. doi: 10.1007/s10120-011-0041-5. No abstract available. PMID 21573743